CLINICAL TRIAL: NCT01014949
Title: Invasive Coronary Microcirculation Assessment in Diabetes and Metabolic Syndrome
Brief Title: Microcirculation Assessment in Diabetes and Metabolic Syndrome
Acronym: MADAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.M. Misericordia Hospital (Other)
Responsible Party: Andrea Picchi, MD, PhD, Interventional Cardiology Unit, Misericordia Hospital, USL 9 Grosseto
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MDM58100
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2009-11

CONDITIONS: Coronary Microvascular Dysfunction; Metabolic Syndrome; Diabetes
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus

ARMS (1):
- Control, Diabetes and Metabolic Syndrome (Other)
  Interventions: Other: Coronary microcirculation assessment

INTERVENTIONS:
Other: Coronary microcirculation assessment — Patients will arrive to the cardiac catheterization laboratory in a fasting state without discontinuation of their cardiac medications. After conventional diagnostic coronary angiography, 3000-5000 I.U. i.v. heparin will be administered, and a 6F coronary guiding catheter will be placed in the ostium of the coronary artery of interest. A 0.014" coronary pressure wire (Radi Medical Systems, Wilmington, Mass) will be calibrated, equalized to the guiding catheter pressure with the sensor positioned in the coronary ostium, and then advanced to the distal coronary artery (down to at least two thirds of the epicardial vessel length). Coronary flow reserve (CFR), fractional flow reserve (FFR) and the index of microvascular resistance (IMR) will be measured after an intravenous infusion of adenosine [140 ug/kg/min] to induce steady state maximal hyperemia.

SUMMARY:
Abnormal coronary microvascular vasodilation has been demonstrated in patients with diabetes and metabolic syndrome, but the role of insulin resistance in its pathogenesis is not clear. The aim of this study is to invasively assess coronary microcirculation and to investigate the relationship of insulin resistance with coronary microvascular dysfunction.

A pressure temperature-sensor-tipped coronary wire will be advanced in coronary arteries without significant lumen reduction. Thermodilution-derived coronary flow reserve (CFR) will be calculated as resting mean transit time (Tmn) divided by hyperemic Tmn (obtained with a 5-min i.v. infusion of adenosine 140 mg/kg/min). An index of microvascular resistance (IMR) will be calculated as the distal coronary pressure at maximal hyperemia divided by the inverse of the hyperemic Tmn. FFR will be calculated by the ratio of Pd/Pa at maximal hyperemia. Insulin resistance (IR) will be assess by the homeostasis model assessment (HOMA) index and plasma IL-6 and TNF-alpha levels will be measured in addition to routine blood examinations before the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable angina or inducible myocardial ischemia
* Coronary arteries without high-grade epicardial stenoses (angiographic stenosis < 50% and fractional flow reserve [FFR] > 0.75)

Exclusion Criteria:

* Significant renal insufficiency (serum creatinine > 1.5 mg/dL), a recent (< 1 week) acute coronary syndrome, heart failure, severe valvular disease, or hypertrophic cardiomyopathy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-11 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Coronary Flow Reserve and Index of Microvascular Resistance values | Outcome measures will be assessed at the end of the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Interventional Cardiology Unit, Misericordia Hospital, Grosseto, Italy

REFERENCES:
- [Derived] Picchi A, Limbruno U, Focardi M, Cortese B, Micheli A, Boschi L, Severi S, De Caterina R. Increased basal coronary blood flow as a cause of reduced coronary flow reserve in diabetic patients. Am J Physiol Heart Circ Physiol. 2011 Dec;301(6):H2279-84. doi: 10.1152/ajpheart.00615.2011. Epub 2011 Oct 7. PMID 21984541